CLINICAL TRIAL: NCT03440957
Title: Osteopathy Treatment for Cancer Pain Related to the Confinement to Bed Pilot Study
Brief Title: Osteopathy Treatment for Cancer Pain Related to the Confinement to Bed
Acronym: OSTEO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 69HCL17_0723
Record Dates: First submitted 2018-02-15; First posted 2018-02-22 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Cancer Patient Confined in the Bed
Keywords: advanced cancer; osteopathy; pain; bedridden
MeSH Terms: conditions — Pain | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteopathy treatment (Other)
  Interventions: Other: Osteopathic treatment

INTERVENTIONS:
Other: Osteopathic treatment — The patients meeting the inclusions criteria will be informed of the study and an osteopathic treatment holistic ,involving all the body will be applied, three time with 2 days between the treatments .Each meeting with the practitioner will last around 40 minutes. The pain and symptoms assessment will be done before and after the treatment .

SUMMARY:
Staying confined in the bed is frequent at the end of life. The cancer patients can also experiment this situation, and consequences are painful, with pain increasing with the time. This pain are related to the joints stiffing , muscles mass decreasing, and tendons retractions . The non pharmacological approach associated with the conventional treatments can be interesting to assess in this frails patients.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman
* Aged 18 years or older
* Having signed informed consent to participate in the study
* Patient affiliated to a social security scheme
* Patient with pain affecting the musculoskeletal system following prolonged bed rest
* Capable to understand French
* Capable of completing self-assessment scales

Exclusion Criteria:

* Patients with bone metastases at risk for the use of osteopathy
* Patients under legal protection measures
* Patients with cognitive impairment preventing self-evaluation
* Patient who is considered too fragile or with a clinical condition too unstable by the doctor refer to be included in the study
* Patients in the pre-agonic or agonic phase

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Decreased pain intensity of 2 points measured by Analog Visual Scale (AVS) before and after the session | 15 days

SECONDARY OUTCOMES:
Decrease in analgesic consumption for pain related to immobilization | 15 days
Decreased 2 points of intensity of other symptoms associated before and after session measured with Edmonton Symptom Assessment System (ESAS). | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Marilène FILBET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France